CLINICAL TRIAL: NCT03618641
Title: Neoadjuvant Phase II Study of TLR9 Agonist CMP-001 in Combination With Nivolumab in Stage IIIB/C/D Melanoma Patients With Clinically Apparent Lymph Node Disease
Brief Title: CMP-001 in Combo With Nivolumab in Stage IIIB/C/D Melanoma Patients With Clinically Apparent Lymph Node Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diwakar Davar (Other)
Collaborators: Checkmate Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Diwakar Davar, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-169
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Melanoma; Lymph Node Cancer
Keywords: Stage IIIB/C/D
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and CMP-001 Combination (Experimental): Prime Phase -Nivolumab 240mg, IV Infusion, every two weeks starting with Cycle 2 ( Cycles 2, 4, 6) for 6 weeks in combination with CMP-001, 5mg, Injection, at Week 1 and the remaining injections, 10 mg will be administered Weeks 2 -7.
  Boost Phase -Nivolumab 240mg, IV Infusion, every two weeks, over a 46 week period in combination with CMP-001, 5mg, administered every 4 weeks for 1 year.
  Interventions: Drug: CMP-001; Biological: Nivolumab

INTERVENTIONS:
Drug: CMP-001 — A molecule comprised of a 30 nucleotide strand, flanked by 10 guanines on either end. The nucleotide strand is surrounded by a Qβ viral-like protein. The intended mechanism of action of CMP-001 in oncology is the activation of TLR9 in pDC within the tumor or the tumor-draining lymph nodes (tumor-associated pDC).
Biological: Nivolumab — A fully human Ig G4 antibody that blocks PD-1. Nivolumab was initially approved by the FDA for the treatment of patients with unresectable or metastatic melanoma and disease progression following ipilimumab and, if BRAF V600 mutation positive, a BRAF inhibitor. Nivolumab has also been FDA approved to treat patients with advanced (metastatic) squamous non-small cell lung cancer (NSCLC) with progression on or after platinum-based chemotherapy, as well as advanced renal cell carcinoma.

SUMMARY:
The purpose this research study is to determine if the combination of nivolumab and CMP-001 improves the likelihood of eradicating (destroying) disease in the lymph node (pathologic response rate).

DETAILED DESCRIPTION:
Patients are being asked to take part in this clinical research study because they have stage IIIB, IIIC or IIID cutaneous (or unknown primary) melanoma with lymph node disease and have yet to undergo surgery. There are two phases, Prime Phase and a Boost Phase. If they participate they will receive nivolumab in combination with CMP-001 for a total of 7 weeks (Prime Phase) prior to surgery. Surgery will be performed approximately 2-4 weeks after completion of the Prime Phase. After recovery from surgery patients will receive additional nivolumab in combination with CMP-001 for approximately 46 additional weeks (Boost Phase).

The main goal of this research study to determine if the combination of nivolumab and CMP-001 improves the likelihood of eradicating (destroying) disease in the lymph node (pathologic response rate). Pathologic responses are associated with improved relapse-free and overall survival in melanoma.

Prior to surgery (Prime Phase) Nivolumab 240mg, will be administered as a 30-minute IV infusion on an outpatient basis. During the Prime Phase, 3 cycles of Nivolumab will be administered every 2 weeks over a 6 week period starting with cycle 2, cycle 4 and then cycle 6.

Prior to surgery (Prime Phase) CMP-001 will be given as an injection from a syringe weekly for a total of 7 weeks. The first injection (week 1), 5mg, will be applied directly into the skin and the remaining injections, 10mg will be administered, will be given intra-tumorally for weeks 2-7.

Surgery will be performed to the cancerous lymph node 2-4 weeks after the Prime Phase is completed.

After recovery from surgery (Boost Phase) Nivolumab will be administered at 240mg every 2 weeks or 480 mg every 4 weeks depending on the physician's preference. CMP-001, 5mg, will be administered by injections intra-tumorally every 4 weeks for up to 54 weeks.

Patients will be followed to assess for survival status until death, withdrawal of consent, or the end of the study, whichever occurs first. This will be done every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the study.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Diagnosis of histologically or cytologically confirmed diagnosis of cutaneous melanoma belonging to one of the following AJCC TNM stages:

   1. Tx or T1-4 and
   2. N1b, or N1c, or N2b, or N2c, or N3b, or N3c and
   3. M0

   Patients are eligible for this trial either at presentation for primary melanoma with concurrent regional nodal and/or in-transit metastasis; or at the time of clinical detected nodal and/or in-transit recurrence; and may belong to any of the following groups:
   * Primary cutaneous melanoma with clinically apparent regional lymph node metastases.
   * Clinically detected recurrent melanoma at the proximal regional lymph node(s) basin.
   * Clinically detected primary cutaneous melanoma involving multiple regional nodal groups.
   * Clinical detected nodal melanoma (if single site) arising from an unknown primary.
   * In-transit and/or satellite metastases with or without regional lymph node involved permitted if considered potentially surgically resectable at baseline.
   * NOTE: Determination of potential resectability must be made at baseline to be eligible for this neoadjuvant study.
   * NOTE: Patients with mucosal and/or uveal melanoma are not permitted to enroll. Patients with melanomas of unknown primary may be enrolled at the discretion of the treating investigator in discussion with Principal Investigator.
4. Presence of injectable and measureable disease based on RECIST 1.1.
5. Willing to undergo tumor biopsy (core, punch, incisional or excisional). Patients must undergo biopsy (core, punch) or open biopsy (incisional, excisional) within 4 weeks of registration on the study.
6. Performance status of 0 or 1 on the ECOG Performance Scale.
7. Demonstrate adequate organ function as defined below performed on screening labs obtained within 4 weeks of registration.

   * Absolute neutrophil count (ANC) ≥1,500 /mcL
   * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L
   * Platelets ≥100,000 / mcL
   * Serum creatinine or Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN.
   * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN.
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN.
   * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
   * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 7 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 26 weeks after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 26 weeks after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. History of uveal or mucosal melanoma.
2. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
   * Note: Subjects with autoimmune disorders of Grade 4 while on prior immunotherapy will be excluded. Subjects who developed autoimmune disorders of Grade ≤ 3 may enroll if the disorder has resolved to Grade ≤1 and the subject has been off systemic steroids at doses >10 mg/d for at least 2 weeks.
5. Active (i.e., symptomatic or growing) central nervous system (CNS) metastases.
6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
7. Has a systemic disease that requires systemic pharmacologic doses of corticosteroids greater than 10mg daily prednisone (or equivalent). Subjects who are currently receiving steroids at a dose of ≤10mg daily do not need to discontinue steroids prior to enrollment Subjects that require topical, ophthalmologic and inhalational steroids would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study. Subjects who require active immunosuppression (greater than steroid dose discussed above) for any reason are excluded.
8. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 26 weeks after the last dose of trial treatment.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137. Prior treatment with ipilimumab or interferon alfa is allowed. Patients with history of allergic or hypersensitivity reaction to interferon alfa or ipilimumab are also excluded.
14. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected. Patients with treated Hepatitis B/C with no evidence of active infection may be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar Davar, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Davar D, Morrison RM, Dzutsev AK, Karunamurthy A, Chauvin JM, Amatore F, Deutsch JS, Das Neves RX, Rodrigues RR, McCulloch JA, Wang H, Hartman DJ, Badger JH, Fernandes MR, Bai Y, Sun J, Cole AM, Aggarwal P, Fang JR, Deitrick C, Bao R, Duvvuri U, Sridharan SS, Kim SW, A Choudry H, Holtzman MP, Pingpank JF, O'Toole JP, DeBlasio R, Jin Y, Ding Q, Gao W, Groetsch C, Pagliano O, Rose A, Urban C, Singh J, Divarkar P, Mauro D, Bobilev D, Wooldridge J, Krieg AM, Fury MG, Whiteaker JR, Zhao L, Paulovich AG, Najjar YG, Luke JJ, Kirkwood JM, Taube JM, Park HJ, Trinchieri G, Zarour HM. Neoadjuvant vidutolimod and nivolumab in high-risk resectable melanoma: A prospective phase II trial. Cancer Cell. 2024 Nov 11;42(11):1898-1918.e12. doi: 10.1016/j.ccell.2024.10.007. Epub 2024 Oct 31. PMID 39486411
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215
- See also: Neoadjuvant vidutolimod and nivolumab in high-risk resectable melanoma: A prospective phase II trial — https://pubmed.ncbi.nlm.nih.gov/39486411/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab and CMP-001 Combination
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All study-eligible patients assigned to treatment arm
Arm/Group | Nivolumab and CMP-001 Combination
Number analyzed (Participants) | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.5 [53 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Disease Stage [Count of Participants; unit: Participants] — Stage III melanoma, also known as regional melanoma, has metastasized (spread) to nearby lymph nodes, lymph vessels, or skin.
  IIIB: tumor is up to 1.0 millimeter thick with or without broken skin (ulceration) or more than 1.0 millimeter and less than 2.0 millimeters IIIC: tumor is up to 2.0 millimeters thick with or without broken skin (ulceration) or more than 2.0 millimeters and less than 4.0 millimeters thick without IIID: tumor is more than 4 millimeters thick with broken skin (ulceration)
  Participants
    Stage IIIB | 15
    Stage IIIC | 16
    Stage IIID | 3

OUTCOME MEASURES:

1. Primary Outcome: Major Pathologic Response Rate (MPR)
Description: Distribution of pathologic response in the 30 evaluable patients. Major pathologic response was defined on surgical specimens analyzed by blinded two independent dermatopathologists using immune related pathologic response criteria (irPRC). Residual viable tumor (RVT) (wherein RVT = viable tumor area/total tumor bed area) was calculated depending on the quantity of viable malignant cells on H&E-stained slides and confirmatory SOX-10-stained representative sections in ambiguous cases; and thresholds defined as follows: complete response (pCR, 0% RVT), major response (pMR, 0%< RVT ≤10%), partial response (pPR, 10%< RVT ≤50%), and pNR (RVT >50%).
Time Frame: Every 6 weeks from start of study treatment, up to 52 weeks
Population: Patients who completed pre-operative therapy and receive surgery were evaluable for MPR; patients who did not undergo surgery for reasons of disease progression precluding surgery (rapid disease progression) were not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and CMP-001 Combination
Number analyzed (Participants) | 30
Participants
  pCR (0% RVT) | 14
  pMR (0%< RVT ≤10%) | 3
  pPR (10%< RVT ≤50) | 3
  pNR (RVT >50%) | 10

2. Secondary Outcome: Radiographic Response Rate
Description: Number of patients with Complete response [CR], partial response [PR], or stable disease [SD], per RECIST v1.1 criteria. Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10mm short axis);PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease [PD], taking as reference the smallest sum diameters while on study. PD: ≥20% (relative) increase in sum of diameters of target lesions referencing smallest sum on study (includes baseline sum if is smallest on study) and, the sum must also demonstrate an absolute increase of at least 5 mm; appearance of one or more new lesions.
Time Frame: Up to 31 months
Population: Treated participants evaluable for radiologic response.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and CMP-001 Combination
Number analyzed (Participants) | 31
Participants
  Partial Response | 14
  Stable Disease | 10
  Progressive Disease | 7

3. Secondary Outcome: Relapse-Free Survival (RFS)
Description: Length of time from the initiation of treatment that patients survive without recurrence of disease. Per RECIST v1.1, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: Up to 31 months
Population: Treated patients evaluable who were radiologically evaluable.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab and CMP-001 Combination
Number analyzed (Participants) | 31
months | NA [22.0 to NA] — Median not reached due to low number of events.

4. Secondary Outcome: 6-month Relapse-free Survival
Description: Percentage of patients who did not experience disease relapse, 6-months post start of treatment.
Time Frame: Up to 6 months
Population: Treated patients evaluable who were radiologically evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab and CMP-001 Combination
Number analyzed (Participants) | 25
percentage of patients | 81 [62 to 91]

5. Secondary Outcome: 12-month Relapse-free Survival
Description: Percentage of patients who did not experience disease relapse, 12 months post treatment.
Time Frame: Up to 12 months
Population: Treated patients evaluable who were radiologically evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab and CMP-001 Combination
Number analyzed (Participants) | 22
percentage of patients | 74 [55 to 86]

6. Secondary Outcome: 24-month Relapse-free Survival
Description: Percentage of patients who did not experience disease relapse, 24-months post start of treatment.
Time Frame: Up to 24 months
Population: Treated patients evaluable who were radiologically evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab and CMP-001 Combination
Number analyzed (Participants) | 12
percentage of patients | 62 [41 to 77]

7. Secondary Outcome: Overall Survival (OS)
Description: The length of time from the start of treatment that patients remain alive.
Time Frame: Up to 31 months
Population: Trial participants remaining alive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab and CMP-001 Combination
Number analyzed (Participants) | 31
months | NA [NA to NA] — Median not reached due to low number of events.

8. Secondary Outcome: 6-month Overall Survival (OS)
Description: Percentage of patients that remain alive.
Time Frame: Up to 6 months
Population: Trial participants remaining alive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab and CMP-001 Combination
Number analyzed (Participants) | 31
percentage of participants | 100 [100 to 100]

9. Secondary Outcome: 12-month Overall Survival (OS)
Description: Percentage of patients that remain alive.
Time Frame: Up to 12 months
Population: Trial participants remaining alive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab and CMP-001 Combination
Number analyzed (Participants) | 27
percentage of participants | 87 [69 to 95]

10. Secondary Outcome: 24-month Overall Survival (OS)
Description: Percentage of patients that remain alive.
Time Frame: Up to 24 months
Population: Trial participants remaining alive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab and CMP-001 Combination
Number analyzed (Participants) | 16
percentage of participants | 83 [63 to 93]

11. Other Pre Specified Outcome: Expression of Inhibitory and Activating Receptors and Ligands
Description: Circulating and intra-tumoral immune cells, including T-cells (CD8, CD4, Tregs) and antigen-presenting cells (monocytes, macrophages, MDSCs), will be compared pre and post nivolumab and CMP-001 combination treatment.
Time Frame: 3 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: TCR Clonality/Diversity Analyses of Circulating and Intra-tumoral CD8+ T-cells
Description: TCR clonality/diversity will be compared pre and post nivolumab and CMP-001 combination treatment.
Time Frame: 3 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Genetic and Transcriptomic Signatures of Response/Non-response
Description: Genetic and transcriptomic signatures will be compared between patients who do and do not respond to study treatment.
Time Frame: 3 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Novel Tumor Imaging Characteristics in Responders and Non-responders
Description: Tumor imaging characteristics will be compared between patients who do and do not respond to study treatment.
Time Frame: 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events monitored up to 31 months, All-Cause Mortality monitored up to 31 months
Description: Adverse Events: Grade 1 and Grade 2 events per CTCAE v4.0 Serious Adverse Events: Grade 3 and Grade 4 events per CTCAE v4.0
Arm/Group | Nivolumab and CMP-001 Combination
All-Cause Mortality (participants affected / at risk) | 9/34
Serious Adverse Events (participants affected / at risk) | 8/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab and CMP-001 Combination (N=34)
Blood and lymphatic system disorders - Other, specifyhypoxemia (Blood and lymphatic system disorders) | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1
General disorders and administration site conditions - Other, specifyBrain Mets (General disorders) | 1
General disorders and administration site conditions - Other, specifyfailure to thrive (General disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Immune system disorders - Other, specifyMyasthenia Gravis (Immune system disorders) | 1
Wound infection (Infections and infestations) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Cardiac troponin I increased (Investigations) | 1
Investigations - Other, specifyinjection site reaction (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifyCellulitis (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures - Other, specifyCraniotomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab and CMP-001 Combination (N=34)
Anemia (Blood and lymphatic system disorders) | 15
Blood and lymphatic system disorders - Other, specifyDecreased Lymphocyte Count (Blood and lymphatic system disorders) | 4
Blood and lymphatic system disorders - Other, specifyDecreased White Blood Cell Count (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specifyPositive D-Dimer (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specifyprolonged PTT (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 3
Cardiac disorders - Other, specifyTachycardia (Cardiac disorders) | 1
Cardiac disorders - Other, specifyTachycardia - Intermittent (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 6
Sinus tachycardia (Cardiac disorders) | 9
Tinnitus (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Endocrine disorders - Other, specifyincreased Free T3 (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 7
Hypothyroidism (Endocrine disorders) | 5
Blurred vision (Eye disorders) | 2
Eye disorders - Other, specifySeeing black spots (Eye disorders) | 1
Flashing lights (Eye disorders) | 1
Floaters (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specifyDecreased Appetite (Gastrointestinal disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 15
Oral pain (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Chills (General disorders) | 23
Edema face (General disorders) | 1
Edema limbs (General disorders) | 6
Fatigue (General disorders) | 18
Fever (General disorders) | 19
Flu like symptoms (General disorders) | 2
General disorders and administration site conditions - Other, specifyCOVID-19 (General disorders) | 1
General disorders and administration site conditions - Other, specifyChest Pain (General disorders) | 1
General disorders and administration site conditions - Other, specifyDecreased appetite (General disorders) | 2
General disorders and administration site conditions - Other, specifyInjection Site Pain (General disorders) | 1
General disorders and administration site conditions - Other, specifyRigors (General disorders) | 4
General disorders and administration site conditions - Other, specifyedema of neck (General disorders) | 1
General disorders and administration site conditions - Other, specifysore throat (General disorders) | 1
General disorders and administration site conditions - Other, specifyswelling at injection (General disorders) | 1
General disorders and administration site conditions - Other, specifyweakness (General disorders) | 1
Infusion related reaction (General disorders) | 3
Injection site reaction (General disorders) | 11
Injection site reactionRigors (General disorders) | 1
Malaise (General disorders) | 1
Neck edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 5
Cytokine release syndrome (Immune system disorders) | 6
Eye infection (Infections and infestations) | 1
Infections and infestations - Other, specifyCellulitis (Infections and infestations) | 1
Infections and infestations - Other, specifyinjection site reaction (Infections and infestations) | 1
Infections and infestations - Other, specifyscalp wound drainage (Infections and infestations) | 1
Infections and infestations - Other, specifytibial infection (Infections and infestations) | 1
Infections and infestations - Other, specifytumor site infection (Infections and infestations) | 1
Infections and infestations - Other, specifywound complications (Infections and infestations) | 1
Joint infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 3
Vaginal infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specifySurgical Site Infection (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specifyinfusion related reaction (Injury, poisoning and procedural complications) | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 7
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 3
Hemoglobin increased (Investigations) | 1
INR increased (Investigations) | 2
Investigations - Other, specifyBUN Increased (Investigations) | 1
Investigations - Other, specifyBlood Lactate Dehydrogenase Increased (Investigations) | 10
Investigations - Other, specifyBlood bilirubin decrease (Investigations) | 1
Investigations - Other, specifyDecreased T4 (Investigations) | 1
Investigations - Other, specifyDecreased protein (Investigations) | 1
Investigations - Other, specifyElevated LDH (Investigations) | 1
Investigations - Other, specifyElevated Platelets (Investigations) | 1
Investigations - Other, specifyFree T4 Increased (Investigations) | 1
Investigations - Other, specifyHypochloremia (Investigations) | 1
Investigations - Other, specifyIncrease Temperature (Investigations) | 1
Investigations - Other, specifyIncreased Free T4 (Investigations) | 1
Investigations - Other, specifyIncreased LDH (Investigations) | 10
Investigations - Other, specifyIncreased Platelets (Investigations) | 1
Investigations - Other, specifyIncreased Prothrombin Time (Investigations) | 1
Investigations - Other, specifyIncreased Uric Acid (Investigations) | 1
Investigations - Other, specifyLDH Increased (Investigations) | 3
Investigations - Other, specifyRight Axilla Pain (Investigations) | 1
Investigations - Other, specifyThyroid Stimulating Hormone Increased (Investigations) | 1
Investigations - Other, specifydecreased TSH (Investigations) | 1
Investigations - Other, specifyincreased BUN (Investigations) | 1
Investigations - Other, specifyincreased Creatinine (Investigations) | 2
Investigations - Other, specifyincreased D dimer (Investigations) | 1
Investigations - Other, specifyincreased INR (Investigations) | 1
Investigations - Other, specifyincreased PT (Investigations) | 1
Investigations - Other, specifyincreased PTT (Investigations) | 1
Investigations - Other, specifyincreased T3 (Investigations) | 1
Investigations - Other, specifyincreased ldh (Investigations) | 2
Investigations - Other, specifyincreased protein (Investigations) | 1
Investigations - Other, specifyincreased temp (Investigations) | 1
Investigations - Other, specifyinjection site swelling (Investigations) | 1
Investigations - Other, specifyplatelet increased (Investigations) | 1
Investigations - Other, specifyrigors (Investigations) | 3
Investigations - Other, specifysoreness at injection site (Investigations) | 1
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 8
Platelet count decreased (Investigations) | 7
Weight gain (Investigations) | 2
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 5
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 7
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 24
Hypophosphatemia (Metabolism and nutrition disorders) | 16
Metabolism and nutrition disorders - Other, specifyIncrease in phosphorus (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specifydecreased appetite (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specifydecreased protein (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specifyhypouricemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specifyloss of appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyIntermittent Back Pain (Musculoskeletal and connective tissue disorders) | 1
Joint Range of Motion Decreased - R Ankle (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyL Ankle Reconstruction (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyLeft hip pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyLeft shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifySpinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyToothache (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyankle injury (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyjoint pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifymuscle cramping in legs (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifymuscle pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyright arm swelling (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifysprained ankle (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Movements involuntary (Nervous system disorders) | 1
Nervous system disorders - Other, specifyRight Facial Drop (Nervous system disorders) | 1
Nervous system disorders - Other, specifyfacial droop - Right Eye (Nervous system disorders) | 1
Nervous system disorders - Other, specifyright sided facial droop (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 5
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 5
Hematuria (Renal and urinary disorders) | 8
Proteinuria (Renal and urinary disorders) | 7
Renal and urinary disorders - Other, specifyFluid Overload (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specifyGlycosuria (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specifyCOPD (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyPneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyhypoxemia (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin and subcutaneous tissue disorders - Other, specifyCellulitis (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifyDry Skin (hands) (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifyRash (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifySquamous Cell (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifyhives (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifymouth/nasal sores (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifyrash at injection site (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifyredness to neck (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifyskin infection (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 2
Hematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 22
Hypotension (Vascular disorders) | 3
Lymphedema (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT03618641/Prot_SAP_001.pdf